CLINICAL TRIAL: NCT02935452
Title: Implementing and Evaluating the GENIE Tool in Southampton Integrated COPD Service: A Clinical Trial to Ascertain Cost Effectiveness and Patient Benefit
Brief Title: Implementing and Evaluating the Genie Tool in COPD
Acronym: GeCop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19175
Record Dates: First submitted 2016-08-25; First posted 2016-10-17 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: COPD; Emphysema
Keywords: Self-management; Supportive self-management; Normalisation process theory; Social networks
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genie (Active Comparator): This group will have the Genie social tool delivered on a one to one basis at discharge points in the study.
  Interventions: Behavioral: GENIE - social networking tool
- Normal Care (No Intervention): This group will have the same questionaires at discharge, but will be offered normal care

INTERVENTIONS:
Behavioral: GENIE - social networking tool — GENIE is a way to help people think about the links they have with others to manage a health problem (local groups, friends, acquaintances, family members, professionals) and to reflect on their involvement in health and wellness activities and their ability to live an ordinary life with a long term condition. By using GENIE and thinking or talking through the GENIE mapping tool, individuals can visualize their network and can reflect on connections that provide value and resources for managing and where there are gaps in support- this might be social, practical or emotional as well as specifically related to a health condition.
  Arms: Genie

SUMMARY:
The Generating Engagement in Network Involvement (GENIE) Tool is designed to support people to find and join social activities in their own neighbourhoods.

Evidence has shown that people with more social support have increased ability to manage long term conditions and ill health.

Patients with Chronic Obstructive Lung Disease (COPD) have difficulty breathing every day; this is both tiring and makes its difficult to socialise as they did prior to having their condition. COPD can be managed with medicines, and exercise, but will never be cured, so it is considered a 'long term condition.'

This study plans to use a social mapping tool (GENIE) with COPD patients that are already part of the community service. The aim of the study is to increase opportunities to socialise and get day to day support outside of the health service.

Patients will be offered either the tool, or usual care.

If the study is successful then use of health care may reduce in the COPD patients already using the COPD service.

DETAILED DESCRIPTION:
The main aim here is to increase long term health care management options in Solent NHS ( National Health Service) Trust by building social capacity to support self-management. The GENIE tool will be introduced into the COPD service to improve options for social groups and exercise when leaving a pulmonary rehabilitation group, or when clinically unable to participate in exercise. The implementation of the GENIE tool aims;

* to build social networking awareness and the importance of utilising existing social resources in the professional and voluntary members of the COPD service
* to use social network mapping techniques and preference elicitation to engage COPD patients in reflecting on their support preferences and needs, help them access further resources and knowledge
* Evaluate the success of the social mapping techniques (GENIE) in the COPD patient population
* Evaluate the cost benefit to the health service of the GENIE in the COPD patient population

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 with a predominant diagnosis of COPD
* Ability to understand spoken English
* Attending PR assessment/ enrolled in Pulmonary Rehabilitation (PR) or maintenance therapy
* Ability and capacity to make their own decision and consent freely

Exclusion Criteria:

* No clear COPD diagnosis
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Ms Welch, Masters, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Welch L, Orlando R, Lin SX, Vassilev I, Rogers A. Findings from a pilot randomised trial of a social network self-management intervention in COPD. BMC Pulm Med. 2020 Jun 8;20(1):162. doi: 10.1186/s12890-020-1130-1. PMID 32513163
- [Result] Bloom I, Welch L, Vassilev I, Rogers A, Jameson K, Cooper C, Robinson S, Baird J. Findings from an exploration of a social network intervention to promote diet quality and health behaviours in older adults with COPD: a feasibility study. Pilot Feasibility Stud. 2020 Feb 6;6:15. doi: 10.1186/s40814-020-0553-z. eCollection 2020. PMID 32042439

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genie | Normal Care
Started | 30 | 30
Completed | 27 | 29
Not Completed | 3 | 1
Not completed — work and life commintment | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genie | Normal Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
FEV1 [Mean (Standard Deviation); unit: litres] | 0.56 (0.23) | 0.51 (0.21) | 0.53 (0.22)
COPD Severity using GOLD Guidelines [Count of Participants; unit: Participants]
  Mild | 8 | 5 | 13
  Moderate | 11 | 9 | 20
  Severe | 7 | 12 | 19
  Very Severe | 4 | 3 | 7
  Unknown | 0 | 1 | 1
Number of people who live with the participant [Count of Participants; unit: Participants]
  1 person live with | 16 | 14 | 30
  2 people live with | 14 | 12 | 26
  3 people or more live with | 0 | 4 | 4
Number of regular visitors for the participants [Count of Participants; unit: Participants]
  no regular visitors | 5 | 9 | 14
  1 - 4 regular visitors | 17 | 9 | 26
  5-10 regular visitors | 6 | 9 | 15
  more than 10 regular visitors | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in EQ ED From Baseline to 3 Months Endpoint
Description: A quality of life indicator, for pre and post Genie in intervention and pre and post usual care. The scale is 0 to 4, the highest quality life is 0, which means the participant has no problem. The reduction means an improvement in life quality of life.
Time Frame: Baseline and change at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genie | Normal Care
Number analyzed (Participants) | 27 | 29
score on a scale | 0.06 (0.21) | 0.04 (0.26)

2. Primary Outcome: Changes in the Symptom Burden of Disease From Baseline to 3 Months
Description: COPD Assessment Tool (CAT) Score, the scale is 0 to 5, 0 is the best score, the participant has no symptoms. The reduction is improvement with the symptoms.
Time Frame: Baseline with change at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genie | Normal Care
Number analyzed (Participants) | 27 | 29
score on a scale | -1.44 (5.91) | -0.14 (6.31)

3. Primary Outcome: Changes in Quality of Life (Mood) From Baseline to 3 Month Endpoint
Description: PHQ-9 ( depression score), the scale is 0 to 27, the best score is 0, which means the participant does not have depression at all. The reduction of the score means an improvement in mood.
Time Frame: Baseline and change at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genie | Normal Care
Number analyzed (Participants) | 27 | 29
score on a scale | -0.69 (5.39) | 0.4 (2.14)

4. Primary Outcome: Changes in Quality of Life (Anxiety) From Baseline to 3 Month Endpoint
Description: GAD-7 (Generalised anxiety score), the scale is 0 to 21, the best score is 0, participants does not have anxiety. The reduction is an improvement in anxiety.
Time Frame: Baseline and change at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genie | Normal Care
Number analyzed (Participants) | 27 | 29
score on a scale | -0.62 (3.89) | 0.76 (3.12)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Genie | Normal Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT02935452/Prot_SAP_000.pdf